CLINICAL TRIAL: NCT07191652
Title: The Association Between Opioid-Free Anesthesia and Postoperative Agitation-Delirium and the Quality of Postoperative Recovery in Pediatric Otolaryngology Cases Monitored With Perioperative Bispectral Index
Brief Title: The Relationship Between Opioid-Free Anesthesia and Postoperative Agitation-Delirium and Quality of Recovery in Pediatric Ear, Nose, and Throat Cases Monitored With Perioperative Bispectral Index
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, İlayda Bilgili Altuntaş, Physician, Istanbul University - Cerrahpasa
Other Study IDs: E-74555795-050.04-1369719
Record Dates: First submitted 2024-09-26; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Ear Throat Nose Surgery; Delirium - Postoperative; Pain Postoperative
Keywords: Opioid-Free Anesthesia; Postoperative Agitation-Delirium; Quality of Postoperative Recovery; Monitored with Perioperative Bispectral Index; ear throat and nose surgery
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opioid Anesthesia: In Group A, according to retrospective patient records, patients who underwent general anesthesia induction with sevoflurane or intravenous propofol, fentanyl, and rocuronium, and whose anesthesia was maintained with sevoflurane and a remifentanil infusion titrated according to BIS monitoring, were included. Perioperative data-including anesthesia induction details, administered drugs and their dosages, and hemodynamic parameters-will be obtained from anesthesia monitoring records.
  Pain and agitation scores will be assessed using the FLACC or NRS and PAED scales, which are routinely applied in the pediatric recovery unit, and these data will be extracted from patient records. Late postoperative pain and patient satisfaction will be evaluated based on follow-up data recorded during routine postoperative outpatient clinic visits.
- Opioid-free Anesthesia: In Group B, according to retrospective patient records, patients who underwent general anesthesia induction with intravenous propofol or sevoflurane, magnesium sulfate, lidocaine, and rocuronium, and whose anesthesia was maintained with magnesium sulfate, lidocaine, dexmedetomidine, and sevoflurane-titrated according to BIS monitoring-were included. Perioperative data, including anesthesia induction details, administered drugs and their dosages, as well as hemodynamic parameters, will be obtained from anesthesia monitoring records.
  Pain and agitation scores will be assessed using the FLACC or NRS and PAED scales, which are routinely applied in the pediatric recovery unit, and these data will be retrieved from patient records.Late postoperative pain and patient satisfaction will be evaluated based on follow-up data recorded during routine postoperative outpatient clinic visits.

SUMMARY:
Delirium is a postoperative complication that hinders a child's recovery and presents challenges in assessment and management. Ear nose throat (ENT) procedures have been suggested as a risk factor for delirium[1]. While numerous studies have explored the effect of sevoflurane on increasing delirium[2], data regarding opioids remain unclear. This study aims to retrospectively evaluate the incidence of emergence agitation and delirium in pediatric patients following otolaryngology surgery under opioid and opioid-free anesthesia approaches that are routinely used in anesthetic practice for these procedures.

Investigators hypothesis posits that a reduced incidence of burst suppression and opioid-free anesthesia may prevent delirium. The primary aim of this study is to retrospectively evaluate the incidence of emergence agitation and delirium following routine opioid-based and opioid-free anesthesia approaches in pediatric patients undergoing ENT surgeries. The secondary aim is to retrospectively assess late postoperative pain and patient satisfaction.

DETAILED DESCRIPTION:
It has been suggested that ear, nose, and throat (ENT) surgeries may be a risk factor for the development of delirium.

This study will be conducted retrospectively following approval from the Ethics Committee, by reviewing the medical records of pediatric patients who underwent ENT surgery at Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Department of Otorhinolaryngology between January 2024 and June 2025. In our clinic, both opioid-restricted and non-restricted general anesthesia techniques are routinely applied in pediatric ENT surgeries, and the data of these patients will be analyzed retrospectively.

Opioid-based and opioid-free anesthesia techniques are routinely employed in pediatric ENT procedures in our institution. This study aims to retrospectively evaluate the incidence of emergence agitation and delirium associated with these different anesthesia approaches.

For patients in both groups, the following data will be extracted from medical records: age, sex, weight, diagnosis, comorbidities, presence of allergies, type and duration of surgery, anesthesia technique (opioid-based or opioid-free), frequency and duration of hypotension based on age-specific mean arterial pressure percentiles, total amount of opioids used or total lidocaine dose, BIS suppression time, average BIS value, requirement for additional analgesics during recovery, time from discontinuation of inhalational agents to extubation, and length of stay in the recovery room.

In the postoperative period, all patients are routinely assessed in the recovery unit using PAED, PONV, and either FLACC or NRS scores, which will be retrieved from patient records. Late postoperative pain and patient satisfaction will be assessed based on data obtained from routine surgical outpatient follow-ups.

Patients aged 2 to 18 years with an ASA physical status of I-II will be included in the study. Patients with liver failure, renal failure, advanced heart block (second or third degree), history of cerebrovascular events, regular opioid use, will be excluded.

The primary objective of this study is to retrospectively evaluate the incidence of emergence agitation and delirium following routinely applied opioid-based and opioid-free anesthesia techniques in pediatric patients undergoing ENT surgery. The secondary objective is to retrospectively assess late postoperative pain and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:The study will include 126 patients

* Aged 2-18 years
* ASA I-II
* Undergoing elective tonsillectomy, adeoidectomy, cochlear implant surgery under general anesthesia.

Exclusion Criteria:

* Patients with ASA 3,4, 5, or 6
* Liver failure
* Advanced heart block (second and third degree)
* Acute cerebrovascular events
* Mental retardation
* Patients with tracheostomy
* Those unwilling to participate

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of 126 pediatric patients aged between 2 and 18 years, who are classified as ASA physical status I or II and are scheduled to undergo elective ear, nose, and throat (ENT) surgery under general anesthesia. These patients will be included based on the eligibility criteria and will be evaluated retrospectively. Patients will be excluded from the study if they fall under ASA classifications III, IV, V, or VI, or if they have a diagnosis of liver failure, advanced heart block (second or third degree), acute cerebrovascular events, mental retardation, or have a tracheostomy. Additionally, any patient or guardian who declines participation will also be excluded.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
WATCHA Score | 1 hour
  The primary aim of the study is to measured the effects of opioid-based versus opioid-free anesthesia procedures on agitation and delirium with WATCHA score(The WATCHA scale has 5 levels: 0-asleep, 1-calm, 2-crying but can be controlled, 3-crying that cannot be controlled and 4-agitated and trashing around) in the postoperative recovery period in children undergoing Ear, Nose, and Throat (ENT) surgeries.
Pediatric Agitation and Delirium Scale | 1 hour
  The primary aim is to assess postoperative agitation scores with Pediatric Agitation and Delirium Scale( all items are scored on a 0-4 point scale as occuring not at all, just a little, quite a bit, very much, or extremely) in the postoperative recovery period in children undergoing Ear, Nose, and Throat (ENT) surgeries.
WATCHA score | 15th minutes
  The primary aim of the study is to measured the effects of opioid-based versus opioid-free anesthesia procedures on agitation and delirium with WATCHA score(The WATCHA scale has 5 levels: 0-asleep, 1-calm, 2-crying but can be controlled, 3-crying that cannot be controlled and 4-agitated and trashing around) in the postoperative recovery period in children undergoing Ear, Nose, and Throat (ENT) surgeries.
Pediatric Agitation and Delirium Scale | 15th minutes
  The primary aim is to assess postoperative agitation scores with Pediatric Agitation and Delirium Scale( all items are scored on a 0-4 point scale as occuring not at all, just a little, quite a bit, very much, or extremely) in the postoperative recovery period in children undergoing Ear, Nose, and Throat (ENT) surgeries.

SECONDARY OUTCOMES:
FLACC | 1 hour
  The secondary aim is to assess postoperative pain scores with NRS or FLACC score(0 to 10 point, with zero meaning "no pain" and 10 meaning "the worst pain imaginable") at 1 hour
FLACC | 15th minutes
  The secondary aim is to assess postoperative pain scores with NRS or FLACC score(0 to 10 point, with zero meanin "no pain" and 10 meaning "the worst pain imaginable") at 1 mounth
Postoperative quality of recovery | 1 month
  The secondary aim is to assess postoperative quality of recovery score (QoR-15- 0 to 150 point, with zero meaning "the worst recovery point" and 150 meaning "the best recovery point") at 1 mounth
Quality of Recovery Score | 1ST week
  The secondary aim is to assess postoperative quality of recovery score (QoR-15- 0 to 150 point, with zero meaning "the worst recovery point" and 150 meaning "the best recovery point") at 1st week
NRS | 15th minutes
  The secondary aim is to assess postoperative pain scores with NRS or FLACC score(0 to 10 point, with zero meaning "no pain" and 10 meaning "the worst pain imaginable") at 1 hour
NRS | 1st hour
  The secondary aim is to assess postoperative pain scores with NRS or FLACC score(0 to 10 point, with zero meaning "no pain" and 10 meaning "the worst pain imaginable") at 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Ç Tütüncü, Professor, Study Director — Istanbul Univerisity-Cerrahpasa Cerrahpasa Faculty of Medicine; Pınat Kendigelen, associate professor, Study Chair — Istanbul Univerisity-Cerrahpasa Cerrahpasa Faculty of Medicine; İlayda Bilgili Altuntaş, Physician, Principal Investigator — Istanbul Univerisity-Cerrahpasa Cerrahpasa Faculty of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vlajkovic GP, Sindjelic RP. Emergence delirium in children: many questions, few answers. Anesth Analg. 2007 Jan;104(1):84-91. doi: 10.1213/01.ane.0000250914.91881.a8. PMID 17179249
- [Background] Yang X, Lin C, Chen S, Huang Y, Cheng Q, Yao Y. Remimazolam for the Prevention of Emergence Delirium in Children Following Tonsillectomy and Adenoidectomy Under Sevoflurane Anesthesia: A Randomized Controlled Study. Drug Des Devel Ther. 2022 Sep 30;16:3413-3420. doi: 10.2147/DDDT.S381611. eCollection 2022. PMID 36203819
- See also: Remimazolam for the Prevention of Emergence Delirium in Children Following Tonsillectomy and Adenoidectomy Under Sevoflurane Anesthesia: A Randomized Controlled Study — https://www.dovepress.com/remimazolam-for-the-prevention-of-emergence-delirium-in-children-follo-peer-reviewed-fulltext-article-DDDT
- See also: Emergence delirium in children: many questions, few answers — https://journals.lww.com/anesthesia-analgesia/fulltext/2007/01000/emergence_delirium_in_children__many_questions,.18.aspx